CLINICAL TRIAL: NCT06513143
Title: Metaverse Surgical Simulation Platform
Acronym: Metaverse
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202305019RINC
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Virtual Reality
Keywords: virtual reality (VR); metaverse; digital twins; simulated surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Virtual reality surgery: The investigators have completed the translation of personalized 3D models from CT images into virtual 3D models displayed on VR glasses using Synapse (Fujifilm). Additionally, the investigators can illustrate reference CT scans, chart summaries, laboratory data, and other medical information within the VR environment.
  Interventions: Other: CT images into virtual 3D model demonstration

INTERVENTIONS:
Other: CT images into virtual 3D model demonstration — The investigators have finished is personalized 3D model translation from CT images into virtual 3D model demonstrated in VR glasses using Synapse.

SUMMARY:
This project aims to combine virtual reality (VR) technologies to construct a metaverse simulation lung surgery platform, which can not only be used as equipment for training novices, but also as a simulated rehearsal before actual surgery, to improve the safety and smoothness of difficult surgeries.

DETAILED DESCRIPTION:
During the training process of surgeons, hands-on operation has always been the highest guiding principle. Even the most basic and simple surgery requires actual operation before it can be truly learned. However, today, with the increasing awareness of patients, it is slowly becoming unfeasible to let novices directly use patients as practice subjects. In addition to being subject to medical ethics, patients are increasingly unwilling to act as guinea pigs for novice surgeons to practice on, so the time it takes for surgeons to mature their surgical skills is getting longer and longer. The metaverse simulation surgery training platform that this project aims to create hopes to train novices through maximized simulation, feedback on hand feel and force, coordination of instruments and other essentials of mature surgeons.

Currently, when the investigators face difficult surgeries, the investigators have many preoperative simulation images (such as Fujifilm's Synapse, Figure 1), as well as intraoperative navigation technology to guide the surgery through the reconstructed physiological structure map. To a certain extent, this is also the prototype of the metaverse surgery platform, but the investigators can do better. Because these simulation tools are currently only auxiliary in nature, such as constructing visible 3D images to let us know the location of the tumor and the relative position of important neighboring organs. In the end, the investigators still have to simulate these auxiliary images in our brains. Not only is there no actual operation, but due to the different experiences of each surgeon, the results of "brain simulation" will also be different. Therefore, such simulations lack reproducibility and are not completely objective. Therefore, the investigators are trying to create a metaverse simulation surgery system so that preoperative simulations and rehearsals can have the greatest degree of realism, precision and objectivity.

ELIGIBILITY:
Inclusion Criteria:

1. Physicians assess suitable candidates.
2. Consent to the use of their high-resolution computed tomography (CT) scan results as digital simulation material for the establishment of a virtual reality surgical platform.

Exclusion Criteria:

1. Those without high-resolution computed tomography (CT) scan results.
2. Any conditions and circumstances that the trial principal investigator believes may affect the establishment of the trial platform.
3. Those who have concerns about providing their own CT data.
4. (For trial user) The exclusion criteria are:

   * (1) Individuals under the age of 18 are excluded.
   * (2) Any condition or circumstance that the principal investigator deems may affect the establishment of the trial platform.
   * (3) Those who have concerns about providing their own data related to using the surgical simulation platform.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed by surgeons with the following conditions will be included in the eligible group:
  1. Complex thoracic surgery,
  2. Large mediastinal tumors,
  3. Interpulmonary tumors,
  4. Patients requiring tracheal transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
questionnaires | Through study completion, an average of 1 year.
  To evaluate the satisfaction levels of students or operators

CONTACTS AND LOCATIONS:
Overall Officials: Xu-Heng Chiang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Surgery, National Taiwain University Hospital, Taipei, Taiwan